CLINICAL TRIAL: NCT06393569
Title: Experience of Security Having Access to Specialized Palliative Care Clinic
Brief Title: Sense of Security With Access to Palliative Outpatient Clinic
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-02274-01
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Access to Specialized palliative outpatient clinic: Patients who have had access to specialized palliative outpatient clinic before admitted to ASiH

SUMMARY:
The aim of the study is to evaluate experience of security, accessibility, and avoidable utilization of health care services in patients who have had access to specialized palliative care clinic (SPCC) compared to those who have not, and to evaluate the relatives' experience of the care.

DETAILED DESCRIPTION:
Palliative care aims to improve the quality of life for patients and families who are affected life-threatening, incurable disease. The concept of palliative care has changed over time and is not longer reserved for patients in the dying phase. More, and more studies show that early integration of palliative care and disease-specific care give positive results. Specifically, palliative care is about prevent and alleviate suffering by early detection of symptoms and treatment of physical, psychological, social and existential problems. In order to provide the best care, a holistic approach is required that takes up what is important right now for the patient, and not focus on only the diagnoses. The care should be person-centred, but it is not entirely clear how this is best achieved.

In an initiative for person-centered care, Palliative care and ASIH, Region Skåne, was the first region in the Sweden to established a new form of care; 'Palliative specialist outpatient clinic' (which was done in 2021). This initiative is a way to support patients who are still receiving disease-specific treatment at their home clinic, which are not specialized in the palliative care needs that may arise. At the same time, the patients do not have that great care needs that they need to be enrolled in specialized palliative care 24/7.

Patients are invited to the study in connection with enrollment at ASiH. All patients who are referred from Palliative specialist reception are consecutively asked about participation in the study. For each patient who previously had contact with the Palliative Specialist Clinic, a patient referred directly from disease-specific care/primary care will be included as to the control group.

Data collection will take place through a self-developed questionnaire where the patient is asked about his experience of security and accessibility in the last 3 months before enrollment in ASiH. Survey questions about safety and accessibility have been chosen as far as possible from among validated questionnaires. If the patient agrees, relatives will also be invited to answer a similar questionnaire. Data on health care consumption, diagnoses and symptoms are collected through Region Skåne's Vårddatabaser and journal review.

ELIGIBILITY:
Inclusion Criteria:

- Patients admitted to included ASiH-unit

Exclusion Criteria:

* Patients with cognitive impairment
* Patients who cannot fill in a questionnaire in Swedish, Arabic or Serbo-Croatian.

Ages: 18 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have hade access to specialized palliative outpatient clinic. As a control group patients who not have had contact with specialized palliative outpatient clinic woill be included.
  Patients with all kind of diagnoses and symtoms that require care at ASiH and specialized palliative outpatient clinic can be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-14 (Actual); Primary Completion 2027-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Experience of security and continuity | 3 months
  Likert scale, 5-point scale where a higher value indicates higher sense of security and continuity.

SECONDARY OUTCOMES:
Avoidable care consumption | 3 months
  Actual number of avoidable contacts with health care system (e.g., emergency department). Data will be collected by Region Skånes Vårddatabaser
Readmissions to hospital. | 3 months
  Actual numbers of readmission. Data will be collected by Region Skånes Vårddatabaser

CONTACTS AND LOCATIONS:
Overall Officials: Maria Schelin, ass.prof, Principal Investigator — Region Skåne
Locations (1):
- ASiH och palliativ vård Skåne, Lund, Sweden